CLINICAL TRIAL: NCT02990364
Title: Analgesia for Neonatal Circumcision: A Randomized Controlled Clinical Trial of EMLA Versus Combination of EMLA, Sucrose and Dorsal Penile Nerve Block or Ring Block
Brief Title: Combination Analgesia for Neonatal Circumcision
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Rana Sharara, Assistant Professor of Pediatrics and Pediatric Critical Care, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SUR.YE.01
Record Dates: First submitted 2016-12-06; First posted 2016-12-13 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Analgesia
Keywords: Circumcision; Analgesia; Controlled Clinical Trial
MeSH Terms: conditions — Agnosia | interventions — Sucrose; Lidocaine; Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control: EMLA Topical Product (Active Comparator): This represents the control group and it is the traditional analgesic used for circumcisions.
  EMLA cream is a eutectic mixture of 2.5% lidocaine and 2.5% prilocaine, used as a topical anaesthetic to diminish pain from cutaneous procedures. Seventy minutes prior to circumcision, the newborn will be placed in the circumcision mold with the legs restrained, and attached to a monitor. 1 gram of EMLA cream will be applied by the nurse to the penis using a syringe and then wrapped with a dressing (Tegaderm). After sixty minutes the Tegaderm and drug will be removed, and the infant will be left to settle until the circumcision.
  Interventions: Drug: EMLA Topical Product
- EMLA + Sucrose (Active Comparator): There is high-quality evidence for the beneficial effect of sucrose (24%) with non-nutritive sucking (pacifier dipped in sucrose) or 0.5 mL of sucrose orally in preterm and term infants. To assess this, 10 ml of sucrose (24%) will be given to the infant during the course of the circumcision.
  In combination to the EMLA cream, the infant will be given sucrose during the circumcision to test the effects of sucrose and sucking on pain management.
  Interventions: Drug: Sucrose; Drug: EMLA Topical Product
- EMLA + Sucrose + Ring Block (Active Comparator): Ring block will be done with 1% lidocaine without epinephrine injected in a band around the penis halfway along the shaft. Ten minutes prior to circumcision, the newborn will be placed in the circumcision mold with the legs restrained, and attached to a monitor. A total of 2 mg/kg of 1% lidocaine without epinephrine will be used to perform the ring block and will be injected in a band around the penis. The block will be done by the circumciser.
  In combination with the ring block, EMLA + sucrose will be given during the circumcision.
  Interventions: Drug: Sucrose; Drug: Lidocaine; Drug: EMLA Topical Product
- EMLA + Sucrose + DPNB (Active Comparator): Dorsal penile nerve block (DPNB) will be done with 1% lidocaine without epinephrine injected at two sites at the base of the penis (2 and 10 o'clock). Ten minutes prior to circumcision, the newborn will be placed in the circumcision mold with legs restrained, and attached to a monitor. A total of 2 mg/kg of 1% lidocaine without epinephrine will be used to perform the block, and equal aliquots in milliliters will be injected at the two sites at the base of the penis. The block will be done by the circumciser.
  In combination with the DPNB, EMLA + sucrose will be given during the circumcision.
  Interventions: Drug: Sucrose; Drug: Lidocaine; Drug: EMLA Topical Product

INTERVENTIONS:
Drug: Sucrose — Sucrose was given to three out of the 4 intervention groups, to assess its effectiveness in managing pain during circumcision.
  Other Names: 25% Sucrose
  Arms: EMLA + Sucrose; EMLA + Sucrose + DPNB; EMLA + Sucrose + Ring Block
Drug: Lidocaine — Lidocaine was given as a local anesthetic via Ring and Dorsal Penile Block to two of the intervention groups, in combination with the topical cream EMLA and sucking on sucrose.
  Other Names: Xylocaine and Lignocaine
  Arms: EMLA + Sucrose + DPNB; EMLA + Sucrose + Ring Block
Drug: EMLA Topical Product — EMLA cream will be applied 70 minutes to the circumcision to all participants of the study.
  Other Names: Eutectic Mixture of Local Anesthetics

SUMMARY:
Circumcision is a commonly performed procedure on newborn males. Clear recommendations and/or guidelines for pain control during the procedure do not exist. The purpose of this research is to compare various forms of analgesia to evaluate which is the more effective for pain reduction. The investigators hope that this study can provide definitive guidelines on the best form of analgesia to use during circumcision. It is important that we perform this study to ensure that in the future newborns' pain during circumcision is effectively managed.

DETAILED DESCRIPTION:
Procedure/Interventions/Drugs Several forms of analgesia, including local anesthetic creams or local anesthetics administered by injection, will be compared as methods of pain control during circumcision. All of these analgesics have already been used for intra-operative pain control during circumcision. The drugs that will be used in the study are all local anesthetics of the amino-amide group, and include lidocaine and prilocaine. Because there is no consensus on the best anesthetic for circumcision, the investigators propose a comparative study. Children taking part in this research will be put into groups which are selected by chance. There will be three different groups. One of the groups will serve as a control group, and in the three other groups combinations of anesthetics will be tested. The control group will be receiving the usual anesthetic used in the normal nursery for pain control during circumcision, while the combination groups will be receiving additional anesthetic agents. Randomization to groups will be done using a random sequence generator. The intervention for each patient will then be placed in a sealed envelope, and will be opened by the individual performing the circumcision at the time the procedure is scheduled.

The following interventions will be used:

EMLA Topical Product:

EMLA cream is a eutectic mixture of 2.5% lidocaine and 2.5% prilocaine, used as a topical anaesthetic to diminish pain from cutaneous procedures. Seventy minutes prior to circumcision, the newborn will be placed in the circumcision mold with the legs restrained, and attached to a monitor. 1 gram of EMLA cream will be applied by the nurse to the penis using a syringe and then wrapped with a dressing (Tegaderm). After sixty minutes they will be returned to the circumstrep, reattached to the monitor, and legs will be restrained. The Tegaderm and drug will be removed, and the infant will be left to settle then the circumcision will take place.

Dorsal Penile Nerve Block (DPNB):

Dorsal penile nerve block is an anesthetic technique first described in 1978, and has since then been extensively evaluated in the management of pain during circumcision. DPNB will be done with 1% lidocaine without epinephrine injected at two sites at the base of the penis (2 and 10 o'clock). Ten minutes prior to circumcision, the newborn will be placed in the circumcision mold with legs restrained, and attached to a monitor. A total of 2 mg/kg of 1% lidocaine without epinephrine will be used to perform the block, and equal aliquots in milliliters will be injected at the two sites at the base of the penis. The block will be done by the circumciser. Five minutes after the block the circumcision will be performed.

Ring Block:

Ring block is another anesthetic technique described in the 1990s that has also been examined for pain control during circumcision. Ring block will be done with 1% lidocaine without epinephrine injected in a band around the penis halfway along the shaft. Ten minutes prior to circumcision, the newborn will be placed in the circumcision mold with the legs restrained, and attached to a monitor. A total of 2 mg/kg of 1% lidocaine without epinephrine will be used to perform the ring block and will be injected in a band around the penis. The block will be done by the circumcising physician. Five minutes later the circumcision will be performed.

Intervention groups:

Control group: (1) EMLA Combination Groups: (2) EMLA + Sucrose (3) EMLA + Ring Block + Sucrose; (4) EMLA + Sucrose + DPNB For all groups the same procedures detailed above for EMLA, DPNB, and ring block will be followed depending on patient grouping.

General:

EMLA will be used on all patients.

Videotaping:

In order to ensure that the study is properly blinded, video-taping of the procedure will need to take place. A video camera will be set to capture the infant's face and torso and the monitor, but not the individual performing the circumcision. The videos will be labeled numerically, and not by patient name. Videos will be viewed by two other individuals (not present at the circumcision itself and not responsible for obtaining consent), and a possible third viewer may be required to resolve conflicting opinions. The video tapes will not be seen by any other individual, and will only be for data collection and pain scoring. They will be kept in the possession of the two principal investigators in a locked drawer in their offices at all times. The video tapes will be destroyed after the completion of the study.

Outcomes:

The primary outcome variable will be the pain score. Pain scores consist of behavioral components of the infant such as facial expression, crying, breathing patterns, arm movement, and leg movement. Secondary outcomes will include effects on heart rate, crying time, and oxygen saturation (obtained from the monitor).

Patients' participation can be ended at any time by the investigator. Significant new findings will be conveyed to the parents of the newborn.

Risks

The main risks of participation in the study are:

1. the adverse effects that might result from circumcision itself, such as pain, bleeding, surgical trauma, local infections, and meatal stenosis.
2. adverse effects that may result from drugs, such as allergic reactions
3. adverse effects that might result from specific drug administration technique, EMLA may result in methemoglobinemia and local skin reactions such as blanching, edema, and erythema. DPNB and ring block may result in bruising, bleeding, and hematomas at the injection site.
4. adverse effects if the anesthetic is erroneously injected systemically.

Although the investigators have taken steps to minimize the risks of this study, there may also be unforeseeable risks.The parents may choose to withdraw consent at any time during the study.

Benefits All the anesthetics that will be used in the study have already been shown to play a role in pain reduction during circumcision, however some seem to be more effective than others. The participating child will directly benefit from the study, since his pain will be controlled to some extent during the circumcision procedure. Furthermore, if the study provides conclusive evidence about the most effective method of analgesia, then guidelines can be instituted so that in the future all newborns will have their pain successfully controlled during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term, newborn males with a gestational age of 37 weeks or more admitted to the newborn nursery at the American University of Beirut Medical Center.

Exclusion Criteria:

* Unhealthy, premature males.

Ages: 1 Day to 3 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The Neonatal Infant Pain Scale (NIPS) | During Circumcision, at 1 hour intervals for 4 hours after circumcision and for blinded evaluation
  The Neonatal Pain Scale (NIPS) is a behavioral assessment tool for measurement of pain in preterm and full-term neonates. This can be used to monitor a neonate before, during and, after a painful procedure such as venipuncture. It was developed at the Children's Hospital of eastern Ontario.
  Parameters:
  1. Facial Expression
  2. Cry
  3. Breathing Pattern
  4. Arms
  5. Legs *
  6. State of arousal
  The Legs parameter was removed for this study, as the legs are not shown in the video and are tied to the circumcision table during the operation. Moreover, following the circumcision the infants are tucked in via blankets that restrict leg movement.

SECONDARY OUTCOMES:
Heart Rate | During Circumcision, at 1 hour intervals for 4 hours after circumcision and for blinded evaluation
  Effects on heart rate, measured by beats/minute
Crying Time | During Circumcision, at 1 hour intervals for 4 hours after circumcision and for blinded evaluation
  Crying time, measured in seconds using a stop watch.
Oxygen Saturation | During Circumcision, at 1 hour intervals for 4 hours after circumcision and for blinded evaluation
  Oxygen Saturation measured in percent

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers outside the scope of the approved list by the Institutional Review Board of the American University of Beirut.
  Only aggregate and de-identified data will be shared.